Version # 3.0, Date: 7MAY2021

# UNIFORMED SERVICES UNIVERSITY CONSENT TO PARTICIPATE IN RESEARCH

**Title:** A Randomized, Controlled, Blinded, Study of Internet-guided Cognitive Behavioral Therapy for Insomnia in Military Service Members with History of Traumatic Brain Injury

Principal Investigator: David L. Brody, MD, PhD

You may be eligible to take part in this research study. This form gives you important information about the study.

Please take time to carefully review this information. You should talk to the researchers about the research study and ask them any questions you have. You may also wish to talk to others (for example, your friends, family, or your personal physician) about your potential participation in this research study. You do not have to take part in this study. Participation is voluntary. You may also leave the research study at any time without penalization.

## 1. KEY INFORMATION:

We are providing the following information so that you can decide if you want and agree (consent) to participate in this research study. Your participation is voluntary, that is, you do not have to participate if you don't want to. The goal of this research study is to test a new therapy called eCBT-I (Internet-guided Cognitive Behavioral Therapy for Insomnia). The study tests if eCBT-I can help people who have traumatic brain injury (TBI) and trouble sleeping (insomnia) to sleep better. The duration of this study is 9 weeks. If you agree to take part in the study, you will be asked to answer questions about your insomnia, and related medical conditions, using your Internet and telephone during those 9 weeks. You will need to spend approximately 1-2 hours per week during the 9 weeks that you are participating in the study. Some study participants will receive the eCBT-I therapy that we are testing on the website. Others will receive information about sleep disorders, but not the therapy on the website. This is done so we can test whether the eCBT-I is helpful. However, at the end of the 9 weeks, the people who did not get the eCBT-I will be able to use it, if they wish to. You might see some improvement in your sleep and related medical conditions, but there is no guarantee that you will, since the eCBT-I program is experimental. On the other hand, your sleep and tiredness might get worse. Additionally, there is the risk of unauthorized access to your study records, although we are taking measures to safeguard them. If you do not wish to participate in this research study, other treatments for insomnia are available (such as, in-person therapy, relaxation training, and medications) and you should discuss them with your personal physician.

Your decision will not affect your future care within MHS, Uniformed Services University (USU), or that given by your personal physician. If you decide to take part in this research study, you will be asked to sign this document. Before you sign this document, be sure you understand


what the research study is about in all sections of the consent form, including the risks and possible benefits to you.

Please tell the researchers if you are taking part in another research study.

# 2. WHAT IS THE PURPOSE AND DURATION OF THIS RESEARCH AND WHO WILL TAKE PART?

You are being asked to participate in this research study because you are suffering from insomnia sleep disorder with a history of TBI.

The purpose of this research study is to determine whether a new form of therapy, eCBT-I, is effective for treating insomnia in military service members and veterans with a history of TBI. Traditional in-person therapy with CBT-I has been proven safe and effective in treating insomnia in the general population, although the efficacy of eCBT-I in military service members with history of TBI is unknown. The intervention you receive through eCBT-I will be designed to replicate the intervention you may receive for insomnia through a local therapist, psychiatrist, or psychologist. However, intervention in this study will be conducted in a self-guided format using the Internet.

There will be about 200 people taking part in this Internet-based study based over a period of 2 years. Your participation in the study will last for up to 6 months. Participation in the study requires access to and frequent use of the Internet through a personal computer, tablet, or smartphone. The duration of your activities will vary from 1-2 hours per week, depending on the research activities involved. A detailed schedule and timeline of the commitment can be found in Section 4 of this document.

This study is looking at eCBT-I, which has not been well-studied in military service members and veterans with history of TBI. This means that the intervention in this study is considered experimental for insomnia.

### 3. SCREENING PROCESS TO QUALIFY FOR PARTICIPATION IN THIS STUDY

Before you can take part in this study, you will need to have some tests and provide some information so that the Investigator can confirm that you qualify for the study. This is called the "Screening Process". The Screening Process will be conducted by telephone. Questions will include details of your medical history as well as enrollment questionnaires related to your insomnia and TBI.

### 4. WHAT WILL HAPPEN IF YOU DECIDE TO BE IN THIS RESEARCH?

If you agree to participate in this study, you will be asked to complete research-related activities for a period of about 6 months. The study team may contact you and your provided contacts by phone, email, or text during this period for research-related purposes. Providing contact information for anyone other than yourself is completely voluntary. If additional contact information is provided, no information regarding the study or results will be shared with the


contacts that you provide. Research-related activities include a review of your medical history, behavioral outcome assessments, questionnaires, and intervention follow up. This study will be conducted entirely over the Internet and telephone. Your participation requires reliable and daily access to the Internet through a connected device. Successful completion of research-related activities will require approximately 1-2 hours per week of involvement during the initial intervention period of up to 9 weeks.

You will be randomly assigned to 1 of 2 groups. Randomization is a process like flipping a coin and means you will have a chance of being assigned to either group. If you are assigned to the active intervention group, you will receive eCBT-I following enrollment in the study. You will also have a 1 in 4 chance of being in the control group, also known as a placebo. A placebo is an inactive, harmless substitute, like a sugar pill, that has the same appearance as the active research study intervention but contains no active therapeutic component. If you are assigned as part of the control group, you will do other activities using the Internet and by telephone that differ from the active intervention being tested to compare its effect on sleep. If you are in the control group, you will be offered free open-label intervention with eCBT-I following the completion of your participation in this study. All participants will be given the opportunity to receive eCBT-I and potentially improve their symptoms of insomnia by participating.

This research study is a blinded study. This means you will not know whether you are receiving the active intervention or the control. Some members of the study team will also not know which group you are assigned until you complete the study. In the event of an emergency, there is a way to find out which one you are receiving.

Some research-related activities may be combined or separated into multiple sessions if it is more convenient for you or the study team. Additional details regarding a timeline of your participation and activities are listed in the table and text below.

Effective Date: 2/27/2020

| Time | Activity | Duration to Completion |
|---|---|---|
| Informed Consent | Review and sign Informed Consent | About 30 minutes |
| Baseline (Day 0) | <ul> <li>Complete enrollment, medical history, outcome assessment, and study questionnaire forms by telephone including: collection of name, phone number, physical address, email address, demographic information, and medical history relating to your insomnia and TBI</li> <li>Complete outcome assessments and sleep questions through online portal (10 diaries within 2 weeks)</li> </ul> | About 1 hour About 1 hour of time in total. Occurs over a period of 10- 28 days |
| Intervention<br>Period (Days<br>0-62) | Complete self-paced homework and reading assignments that are specific to your randomized group assignment (active eCBT-I or control group) via online study portal | The intervention period will last between 6 and 9 weeks depending on level of availability and commitment About 1-2 hours per week |
| Post-Intervention<br>Evaluation (Day<br>63) | Complete outcome assessments and questionnaires through online portal | About 1 hour |
| 3-Month Follow-<br>Up Evaluation<br>(Day 163) | Complete outcome assessments and questionnaires through online portal | About 1 hour |
| Open-Label<br>Intervention<br>(Day 180) | Study team telephone call to receive group assignment. If assigned to the control group, you will be offered free access to online eCBT-I for up to 9 weeks. Technical support will be provided. There will be no outcome assessments or interactions. | N/A |

### Informed Consent:

After you first contact the study team expressing your interest in participating, the study team will schedule a phone call with you. During this call, the study team will explain the study objectives, procedures, risks and benefits, and timeline. The study team will then conduct the informed consent process in which your formal authorization for participation is given electronically. Completion of informed consent will require access to the Internet through a connected device during the telephone discussion. As part of this process, you will be asked several basic questions regarding study objectives, risks, and safety practices to ensure your understanding of the commitment being requested of you. You will be given the opportunity to review and ask questions during and after the process. All participant interaction with the study team will be conducted through the Internet or telephone. You will be required to have reliable access to a telephone and the Internet using a connected device.

### Baseline Evaluation (Day 0):

Following the informed consent process, the study team will guide you through completion of forms necessary for enrollment, medical history, outcome assessments,

and study questionnaires. This will include a telephone discussion with the study team.

This call will last about 1 hour. We will collect your name, phone number, physical address, email address, demographic info, and medical history relating to your insomnia and TBI. The email address you provide will be used for your access to the online study portal and email reminders from the portal. After this telephone discussion, you will be requested to access the online study portal website and complete questions regarding your sleep history and insomnia-related symptoms you

 IRB NUMBER: CNRM-02-9662 IRB APPROVAL DATE: 06/28/2021 IRB EXPIRATION DATE: 06/26/2022

(USUHS) IRB 1

CNRM-92-9662


may be experiencing such as fatigue, anxiety, depression, and migraine headaches. You will be asked to spend between 10-28 days completing sleep diaries prior to being granted access to the intervention. This period is self-paced, so the amount of days it takes you to complete is dependent on your participation. If you are unable to complete the required diaries in the specified timeframe, you may be discontinued from the study.

## Intervention Period (Days 0-62):

During the intervention period you will receive active eCBT-I or control group access to the online study portal. There will be self-paced homework and reading assignments to complete that are specific to your group assignment. The intervention period will last between 6 and 9 weeks depending on your level of availability and commitment, requiring about 1-2 hours per week of your involvement. Participation during the intervention period is completed through the Internet. You will complete the assignments at your own pace.

### Post-Intervention Evaluation (Day 63):

After the intervention period, you will be given the same outcome assessments and questionnaires administered during the baseline evaluation.

### 3 Month Follow-Up Evaluation (Day 163):

The long-term follow up evaluation will occur about 3 months after you complete the intervention period. During the long-term follow-up, you will be given the same outcome assessments and questionnaires administered during the baseline evaluation.

### Open-Label Intervention (Day 180):

The study team will contact you and confirm your successful completion of the study. You will be told which study group you were part of, either active eCBT-I intervention or control. If you were assigned to the control group, you will be offered free access to online eCBT-I for a period of 9 weeks. The study team will provide free technical and logistic support during this period, although no additional outcome assessments or interaction will be required of you.

### Information about the study available to you:

Over the course of the study, the research staff may provide study participants with a summary of study progress when available. These updates will not include any specific information about you. We may also send you a copy of any research publications resulting from this study. This will also include a summary of the findings. Additional information about the study status and results will be available on ClinicalTrials.gov. The study team will be available to answer any questions you have

about the results of the study. You will be notified of any findings that may increase the risk of participating or that would change your willingness to participate in the study.

# 5. WHAT ARE THE RISKS OR DISCOMFORTS FROM BEING IN THIS RESEARCH?

There are risks, discomforts, and inconveniences associated with any research study. These deserve careful thought. You should speak with the study investigator if you have any questions.

(USUHS) IRB 1 **IRB NUMBER: CNRM-02-9662 IRB** APPROVAL DATE: 06/28/2021 IRB Effective Date: 2/27/2020

Page **5** of **13** 

**EXPIRATION DATE: 06/26/2022** 

CNRM-92-9662 Version # 3.0, Date: 7MAY2021

The possible risks and discomforts from participating in this research study include increased fatigue and anxiety following a period of mild sleep restriction during eCBT-I intervention.

Some of the questions asked during behavioral assessments are sensitive and personal in nature. Answering these may cause distress. You are free to stop the study assessments and study participation at any time. Review of study assessments may not be completed by the study team immediately; however, a member of the study team will be available for consultation to address guestions and concerns at any time during your participation in the study. If you experience any thoughts or feelings that require an immediate response or action, you may contact the study team during regular business hours or you may contact The Military Crisis Line, part of the Veterans Crisis Line, a free and confidential support line, via telephone, chat, or text at any time, 24/7. The telephone number for the Military Crisis Line is 1-800-273-8255 or visit www.veteranscrisisline.net/get-help/military-crisis-line for more information.

There are also general risks associated with your participation. Whether you are assigned to the intervention or control group, there is the possibility that your insomnia symptoms may worsen. Additionally, although efforts are made to protect your research study records, there is always a risk that someone could get access to the information researchers have stored about you. You

will be assigned a coded study ID that will be used in place of your true name on all data forms. All data for the study will be kept in a locked file cabinet and room or on a protected electronic system with limited personnel access to minimize this risk.

There may be other risks related to participating in this study that we do not yet know about.

If you experience any adverse effects that could be due to the study, that are not immediate, please call the study team at 301-456-5474. Calls will be answered during the next regular business day. Correspondence will typically be answered in the same day. After hours correspondence will be answered within 24 business hours, whenever possible. In the case of an emergency, hang up and call 9-1-1 or your location's appropriate number for emergency services.

### 6. WHAT ARE THE POSSIBLE BENEFITS FROM THIS RESEARCH?:

The possible benefit to you as a research participant in this research study is an

improvement in insomnia and insomnia-related symptoms from eCBT-I intervention. While an improvement in insomnia symptoms is possible, there is no guarantee that you will directly benefit from being in this research study. All participants who do not receive eCBT-I during the study will be offered a free course of eCBT-I following the study.

Clinical research is important to the advancement of medicine. Participation in this research study will also serve to improve medical understanding and potentially benefit other active and veteran service members with similar challenges.

(USUHS) IRB 1 IRB NUMBER: CNRM-02-9662 IRB APPROVAL DATE: 06/28/2021 IRB EXPIRATION DATE: 06/26/2022


Effective Date: 2/27/2020

CNRM-92-9662


### 7. WHAT ARE THE ALTERNATIVES TO TAKING PART IN THIS RESEARCH?

There are other options for treating your insomnia. Alternative therapies or procedures outside the scope of this research study that may be available to you include: medications, relaxation training, stimulus control, and light therapy. You should talk with your personal physician about these options.

Choosing not to participate in this research study is also an option.

There may be other research studies involving experimental interventions that could be helpful to your condition.

### 8. IS THERE COMPENSATION FOR YOUR PARTICIPATION IN THIS RESEARCH?

No, you will not receive any compensation for participating in this study.

### 9. ARE THERE COSTS FOR PARTICIPATING IN THIS RESEARCH?

No, there are no costs to you for taking part in this research study.

# 10. <u>PRINCIPAL INVESTIGATOR</u> (the person(s) responsible for the scientific and technical direction of the study):

David L. Brody, MD, PhD
Professor of Neurology, Uniformed Services University
Director, Center for Neuroscience and Regenerative Medicine
david.brody@usuhs.edu
301-461-1787

### **Associate Investigator:**

J. Kent Werner, MD, PhD LCDR, MC, USN Asst. Professor of Neurology, Uniformed Services University Director of Research, WRNMMC Sleep Disorders Center j.werner@usuhs.edu

# 11. <u>STUDY SPONSOR</u> (the organizations or persons who oversee the study and are responsible for analyzing the study data):

This study is sponsored by the CNRM. The CNRM was created as a research partnership between military treatment facilities in the National Capital Area and the National Institutes of Health (NIH). The CNRM focuses on the diagnosis and treatment of TBI.

## 12. SOURCE OF FUNDING:

(USUHS) IRB 1


IRB NUMBER: CNRM-02-9662 IRB
APPROVAL DATE: 06/28/2021 IRB
EXPIRATION DATE: 06/26/2022

Uniformed Services University

Center for Neuroscience and Regenerative

This study is funded by the CNRM. Medicine

CNRM-92-9662

13. LOCATION OF THE RESEARCH: Version # 3.0, Date: 7MAY2021

# 14. DISCLOSURE OF FINANCIAL INTERESTS AND OTHER PERSONAL <u>ARRANGEMENTS:</u>

The sponsor of this research study has agreed to reimburse USU for some of the costs related to your participation in this study. Reimbursements will include staffing and material expenses for research activities that would not otherwise be performed through standard medical care such as use of information technology and electronic database services.

# 15. WHO WILL SEE MY INFORMATION (PRIVACY) AND HOW WILL IT BE PROTECTED (CONFIDENTIALITY)?

Records of your participation in this research study may only be disclosed in accordance with state and federal law, including the Federal Privacy Act, 5 U.S.C.552a, and its implementing regulations. DD Form 2005, Privacy Act Statement - Military Health Records, contains the Privacy Act Statement for the records. A copy of DD Form 2005 can be given to you upon request, or you can read on-line at:

https://www.esd.whs.mil/Portals/54/Documents/DD/forms/dd/dd2005.pdf

The research team will keep your research records. These records may be looked at by staff from CNRM, USU, the Institutional Review Board (IRB), and the DoD Higher Level Review as part of their duties. These duties include making sure that the research participants are protected. Confidentiality of your records will be protected to the extent possible under existing regulations and laws but cannot be guaranteed.

Representatives of CNRM, USU, DoD, the Henry M. Jackson Foundation (HJF), NIH, and the United States Food and Drug Administration (FDA) may have access to study data for audit purposes.

Procedures will be taken to protect the confidentiality of the data in this study. Upon providing electronic informed consent, you will be assigned a study ID. The study ID will be used to mask your personal information such as name and other identifiable information in research records. A Master List linking your real name with your study ID will be kept in a locked office and file cabinet or in an electronic database located behind a secure firewall. A firewall is a protection or barrier within a computer to protect the information from being viewed by unauthorized people. Only approved study personnel will have access to information that could be used to distinguish or trace an individual's identity. Study collaborators at the University of Virginia (Charlottesville, VA) and Qualtrics (Provo, UT) will have access to study questionnaires, outcomes measures, and sleep diaries but will not have access to information that could potentially identify you other than the email address you provide to the study team. University

 Effective Date: 2/27/2020 (USUHS) IRB 1 IRB NUMBER: CNRM-02-9662 IRB APPROVAL DATE: 06/28/2021 IRB EXPIRATION DATE: 06/26/2022

CNRM-92-9662


of Virginia will be provided your email address for the purpose of providing access to and use of the online portal. This email will only be used for the purposes of participation in this study. If you do not want them to have access to your personal email address, you may create and provide an email address other than your personal email address. Study collaborators will not share this email address or use it to contact you outside of automatic emails generated by the portal for study participation.

Researchers will make every effort to protect your privacy and confidentiality; however, there are always risks of breach of information security and information loss.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of results. You can search this web site at any time.

Complete confidentiality cannot be promised for military personnel, because information regarding your health may be required to be reported to appropriate medical or command authorities to ensure the proper execution of the military mission, including evaluation of fitness for duty.

For this research study, a Department of Health and Human Services (DHHS) Certificate of Confidentiality is in place to protect your privacy such as your name or other identifying information from being disclosed in any civil, criminal, administrative, legislative or other proceedings, whether at the federal, state or local level. The Certificate cannot be used to resist a demand for information from personnel of the U.S. Government that is used for auditing or evaluation of Federally-funded projects or for information that must be disclosed in order to meet the requirements of the Food and Drug Administration (FDA). Further, the researcher is not prevented from disclosure for reporting matters such as family abuse, sexual assault, reportable communicable diseases, a participant's threatened violence to self or others, or as military regulations

may require. You should understand that the Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

By providing electronic informed consent, you also give your permission for information gained from your participation in this research study to be published in literature, discussed for educational purposes, and used generally to further science. You will not be personally identified; all information will be presented as anonymous data.

### **Additional Research Studies**

You may be eligible for other CNRM-funded or CNRM-collaborative studies. If you would like to be referred to these research studies through a CNRM participant referral program, please visit <a href="https://troops.cnrm.nih.gov">https://troops.cnrm.nih.gov</a>. Your participation in this program is voluntary. If you decide to take part, you will be asked to provide some information about yourself and your health, which will be used to determine your eligibility for CNRM-funded and collaborative studies.

Page **9** of **13** 

Effective Date: 2/27/2020

(USUHS) IRB 1 IRB NUMBER: CNRM-02-9662 IRB

APPROVAL DATE: 06/28/2021 IRB EXPIRATION DATE: 06/26/2022

CNRM-92-9662


Please contact CNRM at <u>CNRMstudies@usuhs.edu</u> with any questions that you may have about participating in this referral program.

In addition, you may provide consent for study staff to provide your name and contact information (email, phone number) to the TROOPS staff. Your information will be sent securely and will not be shared with anyone else. This is voluntary. Please indicate your choice below.

With regard to sharing my contact information with TROOPS CNRM investigators and approved study staff:

| YES, I authorize the sharing of my contact information with TROOPS |
|---------------------------------------------------------------------|
| staff NO, I do not authorize sharing of my contact information with |
| TROOPS staff. |

### 16. LONG TERM USE OF DATA

The investigator has requested to save selected data collected from your participation in this research study for possible use in future related research. This data will not contain information that could be used to identify you.

Data collected during study participation that has been de-identified will be shared with the CNRM Informatics Data Repository and may be transferred to the Federal Interagency Traumatic Brain Injury Research (FITBIR) Database. The purpose of the CNRM Informatics Data Repository is to store a large amount of data so that we can learn more about TBI and how to effectively treat people who may have associated

symptoms.

No identifiable information will accompany your data and all identifiable information will be removed. Your data will be coded with a randomly generated code. The data will be stored indefinitely. Dr. David Brody (Principal Investigator) is responsible for your data until they are received at the CNRM Informatics Data Repository. Before sending your data, we will remove your name and identifying information, and will assign the dataset a code. The key to the code will be kept in a separate secure area by the principal investigator. Once your data is in the CNRM Informatics Data Repository, it may be shared with other repositories/databases and with other CNRM investigators as well as investigators outside of CNRM. These investigators will not be able to identify you.

Your data that is stored at the study origination site or at the CNRM Image Processing Core data base at NIH, may be shared with other collaborators and investigators and used for a variety of research purposes that we may not be able to specify at this time. All information that can identify you will be removed before sharing with any investigator or collaborator.

If you wish to remove your data and stop further data use and sharing, please immediately contact the principal investigator enrolling you in this study in writing. The principal investigator will notify the CNRM Informatics Core and your data will be removed from all repositories and destroyed.


Effective Date: 2/27/2020

(USUHS) IRB 1

IRB NUMBER: CNRM-02-9662 IRB APPROVAL DATE: 06/28/2021 IRB EXPIRATION DATE: 06/26/2022

CNRM-92-9662


### 17. VOLUNTARY PARTICIPATION

The decision to take part in this research study is completely voluntary on your part which means you do not have to take part if you do not want to. You may also leave the research study at any time. If you choose not to take part in this research study or if you leave the study before it is finished, there will be no penalty or loss of benefits to which you are otherwise entitled.

You will be informed if significant new findings develop during the course of this research study that may relate to your decision to continue participation.

### 18. WHAT HAPPENS IF I WITHDRAW FROM THIS RESEARCH?

You may withdraw your consent at any time and stop participating in this research study without affecting your eligibility for care or any other benefits to which you are entitled. Should you choose to withdraw, you must notify the study principal investigator in writing. If you withdraw from this research, you should follow up with your personal physician for any additional assistance with your insomnia symptoms.

If you are receiving the intervention as part of this research study, you will no longer be eligible for such research-related intervention. Contact your personal physician for assistance with your insomnia.

Data collected up until the point of withdrawal may be used in data analysis.

The principal investigator of this research study may terminate your participation in this research study at any time if he determines this to be in your best interest, if you are unable to comply with the procedures required, or if you no longer meet eligibility criteria.

## 19. CONTACT INFORMATION:

## Principal Investigator (PI)

The Principal Investigator or a member of the research staff will be available to answer any questions throughout this study.

Principal Investigator: David L. Brody, MD, PhD

Phone: 301-461-1787

Associate Investigator: Kent Werner, Jr., MD PhD

Phone: 301-346-2696

Mailing Address: 6720B Rockledge Drive, Suite 200, Bethesda, MD 20817

# **Study Team**

Phone: 301-456-5474

Email: cnrm-ecbti@usuhs.edu

(USUHS) IRB 1 Page **11** of **13** 

**İRB NUMBER: CNRM-02-9662 IRB** Effective Date: 2/27/2020 APPROVAL DATE: 06/28/2021 IRB

EXPIRATION DATE: 06/26/2022

CNRM-92-9662

Version # 3.0. Date: 7MAY2021

Uniformed Services University Human Research Protection Program (HRPP) Office The Human Research Protection Program Office Point of Contact and/or Human Protections Administrator (HPA) will be available to answer questions or

discuss concerns you may have about this research study.

Human Protections Administrator/HRPP POC: Petrice Longenecker

Phone: 301-295-0814

# Institutional Review Board (IRB) Office

If you have any questions about your rights as a research participant or if you have concerns or complaints about the research study, please contact the IRB Office at:

**Uniformed Services University** Institutional Review Board (IRB) Office 4301 Jones Bridge Road Room A2051 Bethesda, MD 20814 301-319-4730 IF THERE IS ANY PORTION OF THIS DOCUMENT THAT YOU DO NOT

UNDERSTAND. ASK THE INVESTIGATOR BEFORE SIGNING. YOU MAY CONSULT WITH YOUR PERSONAL PHYSICIAN OR LEGAL ADVISOR, IF YOU

WISH.

Effective Date: 2/27/2020

(USUHS) IRB 1 IRB NUMBER: CNRM-02-9662 IRB APPROVAL DATE: 06/28/2021 IRB EXPIRATION DATE: 06/26/2022


CNRM-92-9662


A signed and dated copy of this document will be given to you.

#### SIGNATURE OF PARTICIPANT

Printed Name of Participant

By signing below, I agree that I have been provided time to read the information describing the research study in the consent form. The content and meaning of this information has been explained to me. I have been provided with the opportunity to ask questions. I voluntarily consent to participate in this study.

ask questions. I voluntarily consent to participate in this study.

By signing this form, I have not given up any of my legal rights as a research participant.

□ I agree to take part in the research described in this consent form.

□ I agree that by checking this box and entering my legal name, I am providing an electronic mark that is held to the same standard as a legally binding equivalent of a handwritten signature.

| Participant's Personal Identifying Nonword Date Tim | e |
|---|---|
| SIGNATURE OF INDIVIDUAL ADMINISTERING CONSENT (Can only be signed by an investigator or staff approved to administer consent) | |
| Printed Name of Administering Individual | |
| Signature of Administering Individual Date Time | |
